CLINICAL TRIAL: NCT03472612
Title: Pathophysiology of Obstructive Sleep Apnoea Recurrence During Continuous Positive Airway Pressure Therapy Withdrawal
Brief Title: OSA Recurrence in CPAP Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 237921
Record Dates: First submitted 2018-03-07; First posted 2018-03-21 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: OSA
Keywords: OSA; CPAP; upper airway collapse; neural respiratory drive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP withdrawal (Experimental): Short-term withdrawal of CPAP therapy in moderate to severe OSA (intervention)
  Interventions: Other: CPAP withdrawal

INTERVENTIONS:
Other: CPAP withdrawal — Short-term withdrawal of CPAP therapy in moderate to severe OSA

SUMMARY:
Continuous positive airway pressure (CPAP) therapy is the most effective Treatment for obstructive sleep apnoea (OSA ). However, adherence to CPAP is often limited. There are established and emerging treatment alternatives to CPAP available, however, they are usually less effective than CPAP. To develop novel treatment methods and to predict who will respond to which treatment, the mechanism underlying obstructive sleep apnoea and different patient types should be described. Especially the contribution of the upper airway function and central respiratory control should be studied for this purpose. In a prospective interventional study, patients with OSA effectively treated with CPAP will undergo physiologic measurements during a two week period off CPAP to define the pathophysiological mechanisms associated with OSA recurrence. This knowledge could facilitate individually tailored treatment and improve therapy adherence and patient outcomes.

DETAILED DESCRIPTION:
Obstructive sleep apnoea (OSA) is a highly prevalent sleep-related breathing disorder characterised by a repetitive collapse of the pharynx during sleep, which results in apnoea or hypopnoea associated with oxygen desaturations and arousal from sleep. Continuous positive airway pressure (CPAP) is the gold standard treatment. Treatment success depends on regular CPAP usage. However, low adherence to CPAP is a frequent problem. It has recently been shown that OSA does not re-occur immediately in all OSA patients upon CPAP therapy withdrawal and that there are different patterns of recurrence of OSA as indicated by repeated sleep studies. So far, the mechanisms of OSA recurrence upon CPAP therapy withdrawal are incompletely understood. Upper airway collapsibility and neuromuscular tone, pharyngeal oedema and inflammation, neural respiratory drive, sleep stage and position may play a role.

In a prospective interventional study, patients with OSA effectively treated with CPAP will undergo physiologic measurements during a two week period off CPAP to define the pathophysiological mechanisms associated with OSA recurrence. In particular, we will investigate the effects of CPAP withdrawal on neural respiratory drive and upper airway function. Inpatient sleep studies and assessments will be performed at baseline (day 0) on CPAP and at follow-up upon CPAP withdrawal (day 14). At the end of the trial patients will return to their established CPAP therapy.

We hypothesise that CPAP withdrawal results in different patterns of OSA recurrence defined by neural respiratory drive and upper airway function. The aim of the proposed project is to study the mechanisms of OSA recurrence by using a validated CPAP withdrawal model. Knowledge on recurrence patterns and different phenotypes of OSA could facilitate individually tailored treatment of OSA and improved therapy adherence and patient outcomes.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18-80 years. Objectively confirmed OSA with an apnoea-hypopnoea- index (AHI) or an oxygen desaturation index (ODI) of ≥20/h at the time of diagnosis (obstructive events).
* Effectively treated with CPAP for > 6 months (AHI on CPAP < 5/h, CPAP usage > 4 hours/night > 70% of the days).

Exclusion criteria:

* Moderate to severe obstructive (FEV1/FVC < lower limit of normal and FEV1 < 70% predicted) or restrictive lung disease (FVC < 60% predicted).
* Daytime pCO2 > 6 kPa (45 mmHg).
* Central Sleep Apnoea/Cheyne Stokes Respiration. Unstable heart failure, untreated coronary artery disease, severe arterial hypertension (resting blood pressure >180/110 mmHg).
* Co-existing non-respiratory sleep disorder (by history).
* Opioid or sedative use. Alcohol abuse.
* Current professional driver or comparable profession.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in neural respiratory drive (NRD) during sleep upon CPAP therapy withdrawal | 2 weeks
  Electromyography of respiratory muscles as measure of neural respiratory drive

SECONDARY OUTCOMES:
Pharyngeal critical occlusion pressure during sleep (Pcrit) | 2 weeks
  Measures of upper airway collapsibility (cmH2O)
Forced oscillation technique (FOT) | 2 weeks
  Measure of (upper) airway resistance
Negative expiratory pressure (NEP) | 2 weeks
  Measure of (upper) airway resistance and collapsibility (cmH2O)
Pharyngeal oedema | 2 weeks
  Transcervical ultrasound (mm)
Forced expiratory volume in 1 second | 2 weeks
  Spirometry
Forced vital capacity | 2 weeks
  Spirometry
Recurrence pattern of OSA defined by the nightly obstructive respiratory events (apnoea-hypopnoea-index) | 2 weeks
  Polysomnography (events/hour)
Recurrence pattern of OSA defined by the nightly obstructive respiratory events (oxygen desaturation index) | 2 weeks
  Nightly home pulse oximetry (events/hour)
Home and office blood pressure | 2 weeks
  Blood pressure (mmHg)
Home and office heart rate | 2 weeks
  Heart rate (bpm)
Epworth Sleepiness Scale Score (ESS) | 2 weeks
  Questionnaire for subjective sleepiness (Points)
Fatigue Severity Sclae (FSS) | 2 weeks
  Questionnaire for subjective sleepiness (Points)
Stanford Sleepiness Scale (SSS) | 2 weeks
  Questionnaire for subjective sleepiness (Points)
Functional Outcomes of Sleep Questionnaire (FOSQ) | 2 weeks
  Quality of life questionnaire
Association between ODI (recurrence pattern of OSA) and neural respiratory drive (NRD) | 2 weeks
  Multivariate Regression modelling with ODI as dependent variable

OTHER OUTCOMES:
Association between different measures of (upper) airway function, namely Pcrit, FOT, NEP and FEV1/FVC | 2 weeks
  Correlation analyses

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Steier, MD Ph, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No